CLINICAL TRIAL: NCT07349810
Title: Continuous Infusion Pump Versus Single Shot Peripheral Block for Pain Management After Same-day Orthopaedic Surgery
Brief Title: Post Operative Infusion Pump Pain Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Charles Gatt, MD, Chair of the Department of Orthopaedic Surgery at Rutgers Robert Wood Johnson, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2022000405
Record Dates: First submitted 2026-01-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Ropivacaine

STUDY DESIGN:
Intervention Model Description: This study will be a pragmatic, prospective cluster randomized trial, where clusters will formed based on sequential 4 week time increments across the study recruitment period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Post-Operative: Continuous ropivacaine via Ambit pump (Experimental): Postoperatively, infusion pump reservoirs will contain 0.20% ropivacaine and infused via the Ambit pump (8cc/hr for knees, 6cc/hr for shoulders).
  Interventions: Drug: Bupivacaine 0.5% Injectable Solution; Drug: Ropivacaine 0.2% Injectable Solution; Device: ambIT Infusion Pump
- Pre-Operative: Liposomal bupivacaine (Exparel) (Active Comparator): A single-shot of Liposomal Bupivicaine (Exparel) will be administered pre-operatively
  Interventions: Drug: Bupivacaine 0.5% Injectable Solution; Drug: 1.3% liposomal bupivacaine (Exparel)

INTERVENTIONS:
Drug: Bupivacaine 0.5% Injectable Solution — Preoperatively, a nerve block consisting of 0.5% bupivacaine will be given to ALL patients
  * A bolus of 20cc will be used for saphenous nerve blocks for knee surgeries
  * A bolus of 15cc will be used for interscalene nerve blocks for shoulder surgeries
Drug: Ropivacaine 0.2% Injectable Solution — Post-operative continuous infusion
  Arms: Post-Operative: Continuous ropivacaine via Ambit pump
Drug: 1.3% liposomal bupivacaine (Exparel) — Pre-operative infiltrative of 10cc of 1.3% liposomal bupivacaine (Exparel)
  Arms: Pre-Operative: Liposomal bupivacaine (Exparel)
Device: ambIT Infusion Pump — A pain pump provides intermittent delivery of medication to manage post-surgery pain.
  Arms: Post-Operative: Continuous ropivacaine via Ambit pump

SUMMARY:
This study will be a pragmatic, prospective cluster randomized trial, where clusters will formed based on sequential 2 week time increments across the study recruitment period.. Patients 18 years or older undergoing ACL reconstruction, open shoulder labrum or rotator cuff surgery, arthroscopic rotator cuff repair, proximal or distal patellar realignment surgery, open knee arthrotomy cases (i.e. inside out meniscus repair, osteochondral allograft transplantation (OCA), meniscal allograft transplantation (MAT)) at University Center for Ambulatory Surgery, LLC (UOA) will be reviewed for eligibility. Once identified, potential study subjects will be asked whether they are interested in participating in the project. If the patient agrees, the subject will be given the informed consent to read and sign.

Objectives: The primary objective is to compare the effectiveness of postoperative infusion pain pump versus preoperative nerve block in reducing visual analog pain scores/numerical pain rating scale (VAS/NPRS) in the postoperative period. The second objective is to evaluate the requirement of narcotic and non-narcotic analgesic medications between the two groups.

Hypotheses: Use of continuous infusion pain pump or single shot peripheral block will result in similar post-operative pain control after outpatient sports medicine surgical cases.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* ACL reconstruction
* Open shoulder labrum or rotator cuff surgery
* Arthroscopic rotator cuff repair
* Proximal or distal patellar realignment surgery
* Open knee arthrotomy cases - Inside out meniscus repair, OCA, MAT

Exclusion Criteria:

* Age under 18 years
* Body mass index of greater than 40 kg/m2
* American Society of Anesthesiologist class 4 physical status or greater
* History of drug or alcohol abuse
* Chronic opioid use/pain management doctor
* Allergy to bupivacaine, ropivacaine or pharmacologic analogs
* Any coagulation disorders
* Existing nerve injury
* Severe bronchopulmonary disease
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of postoperative infusion pain pump versus preoperative nerve block in reducing visual analog pain scores/numerical pain rating scale (VAS/NPRS) in the postoperative period | Postoperative days 0, 1,2,3,4,7,10, 14
  Compare the effectiveness of postoperative infusion pain pump versus preoperative nerve block in reducing visual analog pain scores/numerical pain rating scale (VAS/NPRS) in the postoperative period. NPRS score difference of approximately 1.5 +/- 1 (approximately 2 points) to detect clinically significant difference in pain score.

SECONDARY OUTCOMES:
Evaluate the requirement of narcotic and non-narcotic analgesic medications between the two groups | Postoperative period through day 14
  use of narcotic and other analgesic pain medication throughout the 14 day postoperative period
Safety Outcomes | Postoperative period through day 14
  Evaluate the rates of catheter site infection, extravasation, pump malfunction

CONTACTS AND LOCATIONS:
Locations (1):
- University Center for Ambulatory Surgery, Somerset, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trail, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.